CLINICAL TRIAL: NCT01369134
Title: Clinical Evaluation of 3M ESPE Adper Easy Bond Self-Etch Adhesive Using a Selective Etch Technique
Brief Title: Clinical Evaluation of a Self-etch Adhesive Using a Selective Etch Technique
Status: Completed | Type: Observational
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-10-014
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Dental Caries
Keywords: self-etch adhesive; selective enamel etching; Adper Easy Bond; Supreme Ultra; Molar and premolar teeth; Adult; Class I and II cavities
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Adper Easy Bond Self-etch dental adhesive — Bonding composite to restore Class I or Class II cavities
  Other Names: self etch adhesive with enamel etch

SUMMARY:
Study hypothesis: Etching the enamel followed by use of a self-etching adhesive on enamel and dentin is as effective as a one-step etch and rinse approach.

DETAILED DESCRIPTION:
There is scant evidence available on the performance of self-etching dental adhesive systems. This study aims to clinically evaluate a self-etch adhesive used either with an extra enamel etching step, or in a self-etch stand alone technique with no extra enamel etch.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* written informed consent
* regular dental attender, can return to clinic for study recalls
* good medical health
* normal saliva flow
* has one or two pairs of back teeth that require a Class I or II restoration of appropriate size
* study teeth that are vital

Exclusion Criteria:

* currently in an evaluation of other dental materials
* an irregular dental attender
* has unacceptable oral hygiene standards
* has chronic periodontitis or rampant caries
* has teeth with signs of periapical pathology
* has history of pulp problems, and/or needs pulp treatment
* women who are pregnant or breast-feeding
* has known allergy to resin composite or latex
* has serious chronic disease requiring hospitalization
* has oral soft tissue pathologies
* takes medications which, in the opinion of the investigator, could interfere with the conduct of the study
* has current or recent history of alcohol or other substance abuse
* is an employee of the sponsor or the study site, or members of their immediate family
* has had any restorative treatment of teeth involved in the study in the last twelve months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dental patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Retention of the Restoration | one year
  Bonded filling still in place

SECONDARY OUTCOMES:
Clinical performance of the study restoration | one year
  Restoration in satisfactory clinical function at one year

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Munoz, DDS, Principal Investigator — Dental Clinic Research Center, School of Dental Medicine, 215 Squire Hall, 3435 Main St, Buffalo, NY 14214
Locations (1):
- School of Dental Medicine, Buffalo, New York, United States